CLINICAL TRIAL: NCT00553072
Title: Magnesium Sulphate in Perinatal Asphyxia: A Randomized Placebo Controlled Trial.
Brief Title: Magnesium Sulphate in Perinatal Asphyxia
Acronym: Magsulf
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr.Mushtaq, Professsor, Sheri Kashmir Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKIMS-001
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2013-11

CONDITIONS: Perinatal Asphyxia , Moderate to Severe HIE
Keywords: Asphyxia; perinatal; magnesium sulphate
MeSH Terms: conditions — Asphyxia | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulphate, neurological outcome (Active Comparator): Magnesium sulphate 250mg/kg after every 24 hours starting within 6 hours from birth
  Interventions: Drug: Magnesium sulphate
- Placebo (Placebo Comparator): Placebo every 24 hours for 3 doses starting from 6 hours after birth
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium sulphate — 250 mg/kg/dose in 1 ml normal saline
  Arms: Magnesium sulphate, neurological outcome
Drug: Normal saline — 1 ml/kg/dose
  Arms: Placebo

SUMMARY:
Magnesium sulphate has been shown to be neuroprotective. The investigators hypothesize that magnesium sulphate infusion given to babies with perinatal asphyxia should improve outcome in the immediate neonatal period.

DETAILED DESCRIPTION:
Magnesium sulphate has a neuroprotective potential as has been shown by many studied in pregnant ladies with eclampsia where it helped neonates also and in mothers with preterm labour where the incidence of cerebral palsy was less. We designed a randomised controlled trial on 40 neonates with severe perinatal asphyxia to see whether it helps in the short term outcome of these neonates.

ELIGIBILITY:
Inclusion Criteria:

* Babies eligible for the study were:

  1. Term or post term
  2. Less than 6 hours of age and had
  3. severe perinatal asphyxia as manifested by any three of the following criteria.

     * History of fetal distress (late deceleration, Loss of beat to beat variability, fetal bradycardia, meconium stained amniotic fluid)
     * Need for immediate neonatal ventilation with bag and mask or through endotracheal intubation for 2 minutes or more after delivery
     * A 5-minute Apgar score of < 6
     * Base deficit 15 mEq/L in cord blood or admission arterial or cord blood pH 4.Moderate to severe encephalopathy

Exclusion Criteria:

* Patients with severe IUGR
* Any condition unrelated to asphyxia
* Maternal prenatal magnesium administration
* Metabolic disorder
* Chromosomal anomalies; and
* Congenital malformations were excluded from the study

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
good short term out come | at discharge
  Death and or abnormal neurological outcome at discharge

SECONDARY OUTCOMES:
abnormal neurological examination and abnormal CT Head | at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mushtaq A Bhat, M.D., Principal Investigator — SKIMS; Dr.Javeed I Bhat, M.D., Study Chair — SKIMS
Locations (1):
- Sheri-Kashmir Institute of Medical Scienceds, Srinagar, Jammu and Kashmir, India

REFERENCES:
- [Derived] Bhat MA, Charoo BA, Bhat JI, Ahmad SM, Ali SW, Mufti MU. Magnesium sulfate in severe perinatal asphyxia: a randomized, placebo-controlled trial. Pediatrics. 2009 May;123(5):e764-9. doi: 10.1542/peds.2007-3642. Epub 2009 Apr 6. PMID 19349375